CLINICAL TRIAL: NCT06816758
Title: Evaluation of Diagnosis and Treatment Methods in Corrosive Esophagitis: Analysis of a 26-Year Experience-Based Algorithm
Brief Title: Evaluation of Diagnosis and Treatment Methods in Corrosive Esophagitis: A 26-Year Experience-Based Algorithm
Status: Completed | Type: Observational
Sponsor: Caner İşevi, MD (Other)
Responsible Party: Sponsor-Investigator, Caner İşevi, MD, Principal Investigator, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Other Study IDs: B.30.2.ODM.0.20.08/800
Record Dates: First submitted 2025-01-27; First posted 2025-02-10 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-01

CONDITIONS: Esophageal Diseases
MeSH Terms: conditions — Esophageal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Routine Care for Corrosive Esophagitis — This is an observational study, so participants are not assigned interventions. However, the study investigates the outcomes of patients diagnosed with corrosive esophagitis who received routine clinical care. The exposure of interest includes diagnostic and treatment procedures such as endoscopic evaluation (Zargar classification), proton pump inhibitors, corticosteroid therapy, and surgical interventions for complications like strictures. The outcomes and clinical data collected reflect routine care practices over 26 years.

SUMMARY:
This study aims to evaluate the diagnosis and treatment methods for corrosive esophagitis based on 26 years of clinical experience. It will retrospectively analyze patient records to identify patterns in clinical outcomes, complications, and the effectiveness of treatment strategies. The study focuses on optimizing patient care by proposing a diagnosis and treatment algorithm that can guide future clinical practices. Data will be collected from hospital archives and electronic health records, covering cases of corrosive esophagitis managed at Ondokuz Mayıs University between 1998 and 2024.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with corrosive esophagitis due to corrosive substance ingestion.
* Hospitalized and treated at Ondokuz Mayıs University Thoracic Surgery Department.
* Patients who underwent clinical, laboratory, and radiological evaluations to confirm the diagnosis.
* Patients who were monitored and met follow-up criteria during their treatment.
* Patients above 18 years of age

Exclusion Criteria:

* Patients under 18 years of age.
* Patients who refused hospitalization or treatment.
* Patients who ingested non-corrosive or non-toxic substances (verified by the Ministry of Health Poison Information Center).
* Patients lost to follow-up or did not complete follow-up requirements.
* Patients with incomplete data during the diagnostic or treatment process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study focuses on patients diagnosed with corrosive esophagitis due to the ingestion of corrosive substances. The population includes individuals aged over 18 years who were hospitalized and treated at Ondokuz Mayıs University Thoracic Surgery Department between 1998 and 2024. The patients underwent clinical, laboratory, and radiological evaluations, and their outcomes were assessed retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Esophageal Stricture, Perforation, and Other Related Complications | Within 1 month after hospital admission
  The number of patients who develop esophageal strictures, perforation, or other complications within 1 month post-admission will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayıs University Faculty of Medicine, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes